CLINICAL TRIAL: NCT03526458
Title: Clinical Trial Evaluating the Efficiency of Holmium Laser Settings on Urinary Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-0252; A539800 (Other: UW Madison); SMPH/UROLOGY (Other: UW Madison); Protocol Version 10/30/2017 (Other: UW Madison)
Record Dates: First submitted 2017-11-14; First posted 2018-05-16 (Actual); Results first posted 2021-08-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2020-08

CONDITIONS: Stone Ureter; Stone;Renal; Surgery
Keywords: Holmium Laser; Laser setting; Stone fragmentation
MeSH Terms: conditions — Ureterolithiasis; Nephrolithiasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Holmium:YAG laser: 0.2J&15Hz (Active Comparator): Patients are assigned to treat stones with 0.2J&15Hz of the holmium laser.
  Interventions: Device: Holmium:YAG laser
- Holmium:YAG laser: 0.8J&15Hz (Experimental): Patients are assigned to treat stones with 0.8J&15Hz of the holmium laser.
  Interventions: Device: Holmium:YAG laser

INTERVENTIONS:
Device: Holmium:YAG laser — Treatment of urolithiasis is commonly done using the holmium:YAG laser as this has been shown to be a safe and effective method of treating a wide variety of stones and is currently considered the standard of care (AUA Guideline Panel on the Surgical Management of Stones)

SUMMARY:
The primary objective of this study is to compare the time to acceptable stone fragmentation during clinical use of the holmium laser when using energy settings 0.2J vs 0.8J. The hypothesis is that holmium laser energy settings 0.8J will require less time than lower energy settings 0.2J for fragmenting urinary stones. The clinical practice is to treat urinary stones until the stone is reduced to fragments ≤ 2 mm in size. This is determined by using the laser fiber which is 273 microns to visually estimate the size of the resultant fragments as described by Patel et al, J Endo 2014. Investigators will standardize the effect of stone size by creating a ratio of stone size to treatment time. In this study, the frequency is set at 15Hz. Thus, the study contains two arms: 0.2J&15Hz, and 0.8J&15Hz. Patients will be randomized into the two groups by the ratio of 1:1.

DETAILED DESCRIPTION:
The only interventions imposed on subjects as a result of this study are (1) pre-procedural randomization to laser lithotripsy with either 0.2J or 0.8J energy setting, and (2) the use of patient information in describing results. All the other activities are part of the routine clinical practice in the department. Participation in the study will not alter the patients' preoperative, or postoperative care. During surgery, patients' stones will be treated in accordance with the routine clinical practice of fragmenting stones into small pieces (<2 mm). All patients enrolled will undergo routine post-operative follow up including clinic appointments and imaging evaluation. Any complications will be recorded, reported, and treated appropriately. A fixed frequency will be used (15Hz). Thus, the study contains two arms: 0.2J&15Hz, and 0.8J&15Hz. Patients will be randomized into the two groups by the ratio of 1:1. A total of 1 clinic visit (i.e., the stone surgery, approximately 5-6 hours, depending on the duration of the surgery) is needed for this study.

The study procedures are:

1. A study team member who is affiliated with the patient's clinical care (e.g., the surgeon) will initially approach the patients who are scheduled laser lithotripsy treatment of urinary stones. (i.e. informed that there's a research study they may be eligible for, and asked if they want to learn more about it).
2. If the patient is interested in the study, a member of the research team will approach him/her for enrollment.
3. Once the consent form is obtained, patients' medical background will be reviewed for inclusion/exclusion criteria. Patients who meet the inclusion criteria will be included in the study; patients who do not meet the inclusion criteria will be excluded.
4. Patients will be randomized to either 0.2J&15Hz or 0.8J&15Hz (randomization ratio 1:1) group.
5. Patients will undergo stone surgeries with the laser setting that they are randomized to. The patient's stone(s) will be treated in accordance with the routine clinical practice of fragmenting stone into small pieces (≤ 2mm). The faculty surgeon (i.e., Dr. Nakada) will perform all surgeries.
6. Fragmentation time as well as other information (total surgery time, complications, stone information, and number of stones treated) is collected.
7. After surgery, the patients will then continue on normal postoperative pathway. Postoperative complications will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age
* Patients with urinary stones who require endoscopic treatment

Exclusion Criteria:

* Patients < 18 years of age
* Pregnant patients
* Pre-menopausal females who have not been on approved birth control for at least 1 month pre-operatively
* Patients with stones known to be refractory to treatment with the holmium laser

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Nakada, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Holmium:YAG Laser: 0.2J&15Hz | Holmium:YAG Laser: 0.8J&15Hz
Started | 20 | 20
Completed | 12 | 15
Not Completed | 8 | 5
Not completed — Surgeries rescheduled or cancelled due to COVID | 2 | 2
Not completed — Stone passed, surgery cancelled | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 2 | 1
Not completed — Lack of equipment | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Holmium:YAG Laser: 0.2J&15Hz | Holmium:YAG Laser: 0.8J&15Hz | Total
Number analyzed (Participants) | 12 | 15 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (15.4) | 55.6 (13.1) | 53.6 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 15 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 15 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 15 | 27

OUTCOME MEASURES:

1. Primary Outcome: Fragmentation Time
Description: The time to fragment a stone into small pieces (≤2 mm, which is our current institutional practice)
Time Frame: up to 6 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Holmium:YAG Laser: 0.2J&15Hz | Holmium:YAG Laser: 0.8J&15Hz
Number analyzed (Participants) | 12 | 15
Minutes | 24.5 (19.2) | 7.9 (3.2)
Statistical Analysis 1: Comparison: Holmium:YAG Laser: 0.2J&15Hz vs Holmium:YAG Laser: 0.8J&15Hz; Test type: Superiority; p = 0.012, t-test, 2 sided; Mean Difference (Final Values) = 16.6, 95% CI 2-sided [4.4 to 28.9], Standard Error of Mean 5.6

2. Secondary Outcome: Total Operative Time
Time Frame: up to 6 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Holmium:YAG Laser: 0.2J&15Hz | Holmium:YAG Laser: 0.8J&15Hz
Number analyzed (Participants) | 12 | 15
Minutes | 75.7 (20.6) | 64.3 (17.2)
Statistical Analysis 1: Comparison: Holmium:YAG Laser: 0.2J&15Hz vs Holmium:YAG Laser: 0.8J&15Hz; Test type: Superiority; p = 0.132, t-test, 2 sided; Mean Difference (Final Values) = 11.3, 95% CI 2-sided [-3.6 to 26.3], Standard Error of Mean 7.3

3. Secondary Outcome: Pre-Operative Stone Size
Description: Pre-operative stone size (on pre-operative CT) will be reported in millimeters.
Time Frame: Retrospective review of health chart at Baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Holmium:YAG Laser: 0.2J&15Hz | Holmium:YAG Laser: 0.8J&15Hz
Number analyzed (Participants) | 12 | 15
mm | 11.2 (5.2) | 9.2 (8.2)
Statistical Analysis 1: Comparison: Holmium:YAG Laser: 0.2J&15Hz vs Holmium:YAG Laser: 0.8J&15Hz; Test type: Superiority; p = 0.654, t-test, 2 sided; Mean Difference (Final Values) = 1.2, 95% CI 2-sided [-4.4 to 6.9], Standard Error of Mean 2.7

4. Secondary Outcome: Number of Participants With Either Ureteral or Renal Location of Urinary Stone
Description: Urinary stone location will be classified as renal or ureter.
Time Frame: up to 6 hours
Measure: Number; unit: Participants
Arm/Group | Holmium:YAG Laser: 0.2J&15Hz | Holmium:YAG Laser: 0.8J&15Hz
Number analyzed (Participants) | 12 | 15
Participants
  Ureteral | 8 | 7
  Renal | 4 | 8
Statistical Analysis 1: Comparison: Holmium:YAG Laser: 0.2J&15Hz vs Holmium:YAG Laser: 0.8J&15Hz; Test type: Superiority; p = 0.299, Chi-squared

5. Secondary Outcome: Number of Participants Treated for Either Single or Multiple Urinary Stones
Time Frame: up to 6 hours
Measure: Number; unit: Participants
Arm/Group | Holmium:YAG Laser: 0.2J&15Hz | Holmium:YAG Laser: 0.8J&15Hz
Number analyzed (Participants) | 12 | 15
Participants
  Single | 8 | 14
  Multiple | 4 | 1
Statistical Analysis 1: Comparison: Holmium:YAG Laser: 0.2J&15Hz vs Holmium:YAG Laser: 0.8J&15Hz; Test type: Superiority; p = 0.076, Chi-squared

6. Secondary Outcome: Density of Urinary Stones
Time Frame: up to 6 hours
Measure: Mean (Standard Deviation); unit: Hounsfield units
Arm/Group | Holmium:YAG Laser: 0.2J&15Hz | Holmium:YAG Laser: 0.8J&15Hz
Number analyzed (Participants) | 12 | 15
Hounsfield units | 935.2 (367.9) | 924.7 (374.5)
Statistical Analysis 1: Comparison: Holmium:YAG Laser: 0.2J&15Hz vs Holmium:YAG Laser: 0.8J&15Hz; Test type: Superiority; p = 0.943, t-test, 2 sided; Mean Difference (Final Values) = 10.4, 95% CI 2-sided [-286 to 306.8], Standard Error of Mean 143.9

7. Secondary Outcome: Number of Participants With Urinary Stone Fragment Size of 1, 2 or 3 mm
Description: Size of fragments created will be assessed using the laser fiber size as a comparison.
Time Frame: up to 6 hours
Measure: Number; unit: Participants
Arm/Group | Holmium:YAG Laser: 0.2J&15Hz | Holmium:YAG Laser: 0.8J&15Hz
Number analyzed (Participants) | 12 | 15
Participants
  1mm | 1 | 5
  2mm | 10 | 10
  3mm | 1 | 0
Statistical Analysis 1: Comparison: Holmium:YAG Laser: 0.2J&15Hz vs Holmium:YAG Laser: 0.8J&15Hz; Test type: Superiority; p = 0.185, Chi-squared

ADVERSE EVENTS:
Time Frame: Within 30 days of the surgery
Arm/Group | Holmium:YAG Laser: 0.2J&15Hz | Holmium:YAG Laser: 0.8J&15Hz
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/15
Other Adverse Events (participants affected / at risk) | 0/12 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT03526458/Prot_SAP_002.pdf
  • Informed Consent Form (2017-09-27): https://cdn.clinicaltrials.gov/large-docs/58/NCT03526458/ICF_003.pdf